CLINICAL TRIAL: NCT03123172
Title: The Validity of Central Venous to Arterial Carbon Dioxide Difference to Predict Adequate Fluid Resuscitation During Living Donor Liver Transplantation
Brief Title: The Validity of Central Venous to Arterial Co2 Difference During Living Donor Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Elayashy Mohamed Ahmed Hassan, clinical professor, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N - 21- 2017
Record Dates: First submitted 2017-03-31; First posted 2017-04-21 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-04

CONDITIONS: Liver Transplantation
Keywords: co2 gap; PPV; resuscitation; liver transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- co2 gap (Other): arterial and central venous blood gases to measure Co2 gap
  Interventions: Diagnostic Test: arterial and central venous blood gases

INTERVENTIONS:
Diagnostic Test: arterial and central venous blood gases — withdrawal of arterial and central venous blood gases to measure Co2 gap

SUMMARY:
Study will be conducted on 20 patients ASA III-IV undergoing orthotopic liver transplantation. Blood samples will be obtained simultaneously from arterial line, pulmonary artery catheter and central venous catheter at 4 specific time points baseline, immediately after insertion of PAC; at the end of the dissection phase; 30 minutes after anhepatic phase; 30 minutes after unclamping. Blood samples will be also obtained whenever PPV is more than 15% and patient will need fluid therapy

DETAILED DESCRIPTION:
The study will include 20 ASA II to IV patients with end-stage liver disease, scheduled for orthotropic liver transplantation between. Induction of anaesthesia will be by using propofol (2mg.kg) IV, fentanyl (1-2μg. kg) IV and atracurium (0.5 mg.kg) IV. Anaesthesia will be maintained with Sevoflurane adjusted between 1-2% in an air ⁄ oxygen mix (FiO2 0.6), fentanyl infusion at 1-2 μg.kg/h and atracurium infusion at 0.5 mg.kg/ h. Mechanical ventilation will be provided by using a Dräger anaesthesia machine (Dräger Primus®, Germany) using a tidal volume of 6-8 ml.kg with the respiratory rate adjusted to maintain the PaCO2 between 4-4.6 kPa and PEEP of 5 cmH2O. All patients will be monitored for five lead ECG, peripheral oxygen saturation, noninvasive and invasive arterial blood pressure, temperature, end-tidal carbon dioxide tension, hourly urinary output, and central venous pressure (CVP). A 7-Fr triple lumen CVP catheter (Arrow International Inc, Reading, PA, USA) will be inserted into the right internal jugular vein. A pulmonary artery catheter (OPTIQ SVO2 ⁄CCO; Abbott Laboratories, North Chicago, IL, USA) will also be inserted into the right internal jugular vein. The pulmonary artery catheter (PAC) will be positioned using wedge pressure and confirmed with fluoroscopy.

All patients will receive 6ml /kg/h Ringer acetate solution as a maintenance intraoperative fluid. If PPV is more than 15%, the patient will be considered as fluid responder and will receive a 250-ml bolus of or albumin 5% to maintain PPV ≤15%. Blood transfusion will be given based on a hemoglobin level (< 7 g/dl). Norepinephrine will be administered if the mean arterial pressure was less than 70 mmHg if systemic vascular resistance was less than 600 dyne/sec/cm5 Epinephrine will be administered if mean arterial blood pressure was less than 70 mm Hg and the cardiac index was less than 2.5 L/min/m2 despite sufficient volume infusion, to maintain a target cardiac index of 2.5-3.0 L/min/m2 Blood samples will be obtained simultaneously from arterial line, pulmonary artery catheter and central venous catheter at 4 specific time points baseline, immediately after insertion of PAC; at the end of the dissection phase; 30 minutes after anhepatic phase; 30 minutes after unclamping. Blood samples will be also obtained whenever PPV is more than 15% and patient will need fluid therapy. Central venous oxygen saturation (ScVO2) will be recorded. Pcv-a CO2 gap will be calculated from a sample taken from the central venous catheter, the tip of which was conﬁrmed to be in the superior vena cava near or at the right atrium by radiography. Mixed venous-arterial carbon dioxide (Pmv-a CO2 gap) will be obtained from tip of pulmonary artery catheter All blood gases measurements will be made using a Cooximeter (ABL 700, Radiometer, Copenhagen, Denmark). Immediately after blood samples withdrawal, mean arterial blood pressure (MAP), heart rate, and cardiac output (CO) and arterial lactate will be recorded. Cardiac output will be determined by thermodilution technique using the PA catheter (Abbott Critical Care Systems, North Chicago).

ELIGIBILITY:
Inclusion Criteria:

* ASA II to IV patients with end-stage liver disease
* patients undergoing orthotopic living donor liver transplantation
* age > 18 years

Exclusion Criteria:

* acute fulminant liver failure
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
correlation between the PPV(pulse pressure variation) and Pcv-a CO2 (central venous to arterial) gap | baseline 5 min after induction of anesthesia, immediately after insertion of PAC; 30 minutes after the dissection phase; 30 minutes after anhepatic phase; 30 minutes after unclamping
  changes in central venous to arterial co2 gap with fluid status

SECONDARY OUTCOMES:
correlation between the PPV(pulse pressure variation) and Pmv-a CO2(mixed venous to arterial) gaps | baseline 5 min after induction of anesthesia, immediately after insertion of PAC; 30 minutes after the dissection phase; 30 minutes after anhepatic phase; 30 minutes after unclamping
  changes in mixed venous to arterial co2 gap with fluid status
validity of venous-arterial CO2 gap to predict fluid Responsiveness. | baseline 5 min after induction of anesthesia, immediately after insertion of PAC; 30 minutes after the dissection phase; 30 minutes after anhepatic phase; 30 minutes after unclamping
  sensitivity and specificity of co2 gap to detect patients who are fluid responder and non responder using area under ROC curve
correlation between the CO and both Pcv-a CO2 and Pmv-a CO2 gaps | baseline 5 min after induction of anesthesia, immediately after insertion of PAC; 30 minutes after the dissection phase; 30 minutes after anhepatic phase; 30 minutes after unclamping
  changes in mixed and central venous to arterial co2 gap with cardiac output changes

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mohamed mokhtar, M.D, Study Director — kasralainy faculty of medicine, Cairo university
Locations (1):
- Kasr Alainy Hospital , Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bechstein WO, Neuhaus P. [Bleeding problems in liver surgery and liver transplantation]. Chirurg. 2000 Apr;71(4):363-8. doi: 10.1007/s001040051066. German. PMID 10840602
- [Background] Donati A, Loggi S, Preiser JC, Orsetti G, Munch C, Gabbanelli V, Pelaia P, Pietropaoli P. Goal-directed intraoperative therapy reduces morbidity and length of hospital stay in high-risk surgical patients. Chest. 2007 Dec;132(6):1817-24. doi: 10.1378/chest.07-0621. Epub 2007 Oct 9. PMID 17925428
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Changes in central venous saturation after major surgery, and association with outcome. Crit Care. 2005;9(6):R694-9. doi: 10.1186/cc3888. Epub 2005 Nov 8. PMID 16356220
- [Derived] ELAyashy M, Hosny H, Hussein A, AbdelAal Ahmed Mahmoud A, Mukhtar A, El-Khateeb A, Wagih M, AboulFetouh F, Abdelaal A, Said H, Abdo M. The validity of central venous to arterial carbon dioxide difference to predict adequate fluid management during living donor liver transplantation. A prospective observational study. BMC Anesthesiol. 2019 Jun 22;19(1):111. doi: 10.1186/s12871-019-0776-9. PMID 31228943